CLINICAL TRIAL: NCT04847271
Title: Implementation of Physical Activity on Prescription for Children With Obesity in Paediatric Health Care (IMPA): a Feasibility Study
Brief Title: Physical Activity on Prescription for Children With Obesity
Acronym: IMPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Susanne Bernhardsson, Principal investigator, Research and Development Strategist, R&D primary health care, Vastra Gotaland Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01244
Record Dates: First submitted 2021-03-29; First posted 2021-04-19 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Childhood
Keywords: obesity, childhood; physical activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity on prescription (Experimental): Physical activity on prescription is a behaviour change intervention comprising 3 components: a person-centred pre-intervention dialogue, a written prescription for individually tailored physical activity, and a structured follow-up.
  Interventions: Behavioral: Physical activity on prescription (PAP)

INTERVENTIONS:
Behavioral: Physical activity on prescription (PAP) — The intervention in this study will comprise the 3 PAP components. Participants will take part in all components and perform one or several physical activities of their choice in accordance to the written prescription, at the prescribed frequency and duration, for a period of 4 months.

SUMMARY:
Background: physical inactivity is a main cause of childhood obesity. Physical activity on prescription (PAP) is an evidence-based intervention for adults, but has not been evaluated in children with obesity.

Aim: to evaluate the feasibility of a PAP intervention for children with obesity by assessing both clinical patient outcomes and implementation outcomes.

Method: a single-arm clinical trial in which children with obesity participate in a 4-month PAP intervention. Measurement points are baseline and 4 months, with long-term follow-ups at 8 and 12 months.

Population: children with obesity.

Intervention: physical activity on prescription (PAP).

Patient outcomes: physical activity level/pattern (including sedentary time), BMI, waist circumference, metabolic risk markers, health-related quality of life, self-efficacy for physical activity, motivation for physical activity.

Implementation outcomes: coherence, cognitive participation, collective action, and reflexive monitoring in relation to PAP (the four core constructs of the Normalization Process Theory); appropriateness, acceptability and feasibility of PAP; barriers and facilitators for implementing PAP; recruitment and attrition rates, and intervention fidelity and adherence.

DETAILED DESCRIPTION:
Physical inactivity is a main cause of childhood obesity which tracks into adulthood obesity, making it important to address early in life. Physical activity on prescription (PAP) is an evidence-based intervention developed in Sweden that has shown good effect on physical activity levels in adults, but has not been evaluated in children with obesity. This clinical study is nested in a larger research project aiming to assess the prerequisites, determinants, and feasibility of implementing PAP adapted to children with obesity in paediatric health care. Children's and parents' experiences of participating in the PAP intervention will also be explored.

In a first, pre-clinical trial, phase, healthcare providers and managers from 26 paediatric clinics in Region Västra Götaland, Sweden, will participate in a web-based survey, and a subset of this sample in a focus group study. Findings from these two data collections will form the basis for further development and adaptation of PAP to the target group and context.

In the project's second phase, this adapted PAP intervention will be evaluated in a clinical study in a sample of approximately 60 children with obesity, between 6 and 12 years of age, and one of their parents/legal guardians. Clinical and implementation outcomes will be assessed pre- and post-intervention, and at 8 and 12 months' follow-up. Clinical outcomes are physical activity level/pattern, BMI, waist circumference, metabolic risk markers (blood pressure, fasting plasma glucose, high- and low-density lipoprotein cholesterol, insulin resistance, and triglycerides), quality of life, self-efficacy and motivation for physical activity, and intervention satisfaction. Implementation outcomes are the four core constructs of the Normalization Process Theory; coherence, cognitive participation, collective action, and reflexive monitoring; appropriateness, acceptability and feasibility of the PAP intervention; barriers and facilitators for implementing PAP; recruitment and attrition rates, and intervention fidelity and adherence.

The clinical study is nested in a larger research project employing a hybrid implementation-effectiveness design. Design and analysis of the included studies is guided by the Normalization Process Theory.

ELIGIBILITY:
Pre-trial phase/healthcare practitioner:

Inclusion criteria:

- being a healthcare practitioner or manager involved in the treatment of children with obesity at a paediatric healthcare clinic in Region Västra Götaland

Clinical trial/patients:

Inclusion criteria:

* aged 6-12 years
* diagnosed with obesity (age adjusted BMI>ISO-BMI 30)
* having an insufficient physical activity level according to national recommendations
* being willing to participate and perform the chosen activity/-ies
* having a parent who is willing to participate.

Exclusion criteria:

* severe psychiatric comorbidity
* severe intellectual or physical disability

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity level | 4, 8, 12 months after baseline
  Change in time spent in moderate to vigorous physical activity, measured with accelerometry

SECONDARY OUTCOMES:
Change in physical activity pattern | 4, 8, 12 months after baseline
  Change in sedentary time, time spent in low, moderate and vigorous physical activity, measured with accelerometry
Change in BMI | 4, 8, 12 months after baseline
  Change in age- and sex adjusted BMI (measured as weight and height combined to BMI). This outcome will also be measured as BMI Standard deviation score (SDS)
Change in health-related quality of life | 4, 8, 12 months after baseline
  Change in self-reported health-related quality of life, measured with KIDSCREEN-10
Change in self-efficacy for physical activity | 4, 8, 12 months after baseline
  Change in perceived self-efficacy for physical activity, measured with the Self-efficacy for physical activity questionnaire
Change in motivation for physical activity | 4, 8, 12 months after baseline
  Change in perceived motivation for physical activity, measured with the Motivation for physical activity questionnaire
Intervention acceptability | Post-intervention at 4 months
  Intervention acceptability will be measured with the Client Satisfaction Questionnaire (CSQ-8)
Change in systolic and diastolic blood pressure | Baseline to 12 months
  Both systolic and diastolic blood pressure will be measured in mmHg
Change in fasting plasma glucose | Baseline to 12 months
  Change in fasting plasma glucose will be measured in mmol/litre
Change in Hemoglobin A1C (HbA1C) | Baseline to 12 months
  Change in HbA1C will be measured in mmol/litre
Change in high- and low-density lipoprotein cholesterol | Baseline to 12 months
  Change in high- and low-density lipoprotein cholesterol will be measured in mmol/litre
Change in fasting P-insulin | Baseline to 12 months
  Change in fasting P-insulin will be measured in mIE/litre
Change in triglycerides | Baseline to 12 months
  Change in triglycerides will be measured in mmol/litre

OTHER OUTCOMES:
Change in healthcare practitioners' attitudes towards PAP in relation to the four core constructs of the NPT: coherence, cognitive participation, collective action, and reflexive monitoring | Pre-implementation to post-intervention at 4 months, and long-term follow-up at 12 months
  Coherence, cognitive participation, collective action, and reflexive monitoring will be assessed using the Swedish version of Normalization MeAsure Development (S-NoMAD)
Change in healthcare practitioners' acceptability of the PAP intervention | Pre-implementation to post-intervention at 4 months, and long-term follow-up at 12 months
  Acceptability of PAP will be assessed using the Acceptability of Intervention Measure (AIM)
Change in healthcare practitioners' appropriateness of the PAP intervention | Pre-implementation to post-intervention at 4 months, and long-term follow-up at 12 months
  Appropriateness of PAP will be assessed using the Intervention Appropriateness Measure (IAM)
Change in healthcare practitioners' feasibility of the PAP intervention | Pre-implementation to post-intervention at 4 months, and long-term follow-up at 12 months
  Feasibility of PAP will be assessed using the Feasibility of Intervention Measure (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bernhardsson, Assoc. Prof., Principal Investigator — Vastra Gotaland Region
Locations (1):
- Regionhälsan, Region Västra Götaland, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request
Time Frame: After completion of the study and publication of study results

REFERENCES:
- [Derived] Bernhardsson S, Boman C, Lundqvist S, Arvidsson D, Borjesson M, Larsson MEH, Lundh H, Melin K, Nilsen P, Lauruschkus K. Implementation of physical activity on prescription for children with obesity in paediatric health care (IMPA): protocol for a feasibility and evaluation study using quantitative and qualitative methods. Pilot Feasibility Stud. 2022 Jun 1;8(1):117. doi: 10.1186/s40814-022-01075-3. PMID 35650617